CLINICAL TRIAL: NCT00809419
Title: A Study of the NeoVista Ophthalmic System for the Treatment of Subfoveal Choroidal Neovascularization Associated With Wet Age-Related Macular Degeneration in Patients That Require Persistent Anti-VEGF Therapy
Brief Title: A Study of the NeoVista Ophthalmic System for the Treatment of Subfoveal CNV Associated With Wet AMD in Patients That Require Persistent Anti-VEGF Therapy
Acronym: MERITAGE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NeoVista (Industry)
Responsible Party: Jeffrey A. Nau, MMS, Director of Clinical Affairs, NeoVista, Inc., Kings College Hospital; London, UK
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NVI-008
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Age Related Macular Degeneration
Keywords: Brachytherapy; EpiRad; Macular Degeneration; Ranibizumab
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): NeoVista Ophthalmic System procedure + Lucentis
  Interventions: Device: NeoVista Ophthalmic System

INTERVENTIONS:
Device: NeoVista Ophthalmic System — A single procedure with the NeoVista Ophthalmic System, with Lucentis (0.5mg) administered on an as needed basis for three years.

SUMMARY:
The objective of the MERITAGE Trial is to evaluate the safety and efficacy of focal delivery of radiation for the treatment of subfoveal choroidal neovascularization (CNV) associated with wet age-related macular degeneration (AMD) in patients that require persistent injections of Anti-VEGF therapy to maintain an adequate response to treatment.

DETAILED DESCRIPTION:
Therapeutic advances in the arena of neovascular age-related macular degeneration (AMD) have provided multiple treatment options for the disease. Brachytherapy has been studied in multiple clinical trials in the past with many studies showing a therapeutic benefit. Treatment with radiotherapy and anti-VEGF compounds is a promising approach to treating AMD. The current treatment for neovascualar AMD involves multiple injections over an indefinite period of time. This trial will evaluate whether treatment with brachytherapy can reduce or eliminate the need for continued injections.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have predominantly classic, minimally classic, or occult with no classic lesions, as determined by the Investigator, secondary to AMD, with a total lesion size (including blood, scarring, and neovascularization) of < 12 total disc areas (21.24 mm2) and a GLD ≤5.4 mm.
* Subjects must have completed anti-VEGF induction treatment, defined as the first 3 months of treatment. Following the induction period, subjects must have required at least 5 additional injections of Avastin or Lucentis in the 12 months preceding enrollment, or 3 additional injections of Avastin or Lucentis in the 6 months preceding enrollment, given on an as needed basis. Subjects may have previously received Macugen, although must meet the criteria above for Lucentis or Avastin.
* Subjects must be age 50 or older

Exclusion Criteria:

* Subjects with prior or concurrent subfoveal CNV therapy with agents, surgery or devices (excluding Macugen, Avastin, or Lucentis) including thermal laser photocoagulation (with or without photographic evidence), photodynamic therapy, intravitreal or subretinal steroids, and transpupillary thermotherapy (TTT)
* Subjects who underwent previous radiation therapy to the eye, head or neck
* Subjects who have been previously diagnosed with Type I or Type II Diabetes Mellitus. Subjects that DO NOT have a documented diagnosis, but have retinal findings consistent with Type I or Type II Diabetes Mellitus.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2008-11; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Number of re-treatment injections of anti-VEGF (Lucentis) therapy | 3 years
Percentage of subjects losing less than 15 ETDRS letters | 3 years
Safety Assessment: Incidence and severity of averse events and ocular AEs. Incidence of cataract changes. Incidence of radiation induced toxicity | 3 years

SECONDARY OUTCOMES:
Percentage of subjects gaining ≥ 15 ETDRS Letters | 3 years
Percentage of subject gaining ≥0 ETDRS letters | 3 years
Mean change in ETDRS visual acuity | 3 years
Change in total lesion size and CNV size by fluorescein angiography | 3 years
Foveal thickness measured using OCT. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Tim Jackson, MD, Study Director — Kings College Hospital
Locations (5):
- United States (2):
  - Retina Consultants of Arizona, Phoenix, Arizona
  - Retinal Institute of Hawaii, Honolulu, Hawaii
- Israel (2):
  - Rabin Medical Center, Petah Tikva
  - Tel-Aviv Medical Center, Tel Aviv
- Kings College Hospital, London, United Kingdom